CLINICAL TRIAL: NCT06122519
Title: Disorders and the Effect of Corresponding Treatment on the Quality of Life of Children and Adolescents With Autism and Their Caregivers
Brief Title: Characteristics of Eye Diseases in Children and Adolescents With Autism Spectrum Disorders and the Effect of Corresponding Treatment on the Quality of Life of Children and Adolescents With Autism and Their Caregivers
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tianjin Eye Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: YK2023002
Record Dates: First submitted 2023-11-03; First posted 2023-11-08 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Autism Spectrum Disorder; Visual Function
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study mainly investigated the incidence of eye diseases in children with autism spectrum disorder(ASD) in Tianjin area, and analyzed related risk factors, so as to raise attention to eye diseases in children with ASD. To evaluate the impact of ophthalmic treatment on the quality of life of children with autism and their primary caregivers.

DETAILED DESCRIPTION:
In recent years, the incidence of autism has increased year by year, which has brought a heavy burden to society and families. For the special group of children with autism spectrum disorder, previous studies focused on the lack of comprehensive and accurate visual function characteristics and defects of this group. In the early stage, it was believed that there was a certain correlation between visual impairment and autism, and some patients with visual impairment were misdiagnosed as autism. Moreover, some studies have shown that the incidence of refractive errors and oblique amblyopia in autistic children is significantly higher than that in normal children. This study mainly includes two parts: On the one hand, investigate the autism children in Tianjin area to understand the incidence of eye diseases. On the other hand, children with eye problems were given relevant interventions, such as optometry, amblyopia training, strabismus surgery, etc., to assess the impact of the corresponding treatment on the quality of life of the children and their primary caregivers.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with ASD but without medical intervention. To cooperate with relevant inspectors.

Exclusion Criteria:

* Brain organic diseases (such as tumors, strokes, epilepsy, etc.) and serious physical diseases (such as heart, liver, kidney and other organ dysfunction, cancer, etc.);Do not cooperate to check.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The plan is to enroll nearly 1,000 children with autism in the study.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
refractive error | 6 months
  Patients with ametropia were given endoscopic treatment, followed up for at least half a year, and the influence of endoscopic treatment on the quality of life of children, adolescents and primary caregivers was observed
strabismus | 6 months
  Patients with strabismus requiring surgical correction were given surgical treatment, followed up for at least half a year, and the effects on the quality of life of children, adolescents and primary caregivers were observed
amblyopia | 6 months
  Patients with amblyopia were treated with amblyopia, followed up for at least half a year, and the influence of the quality of life of children and adolescents and the main caregivers after optometry was observed

SECONDARY OUTCOMES:
OCTA | 6months
  Fundus blood perfusion and retinal thickness were observed
eye tractor | 6months
  The correlation between eye movement and visual function was assessed

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Eye Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided